CLINICAL TRIAL: NCT05300022
Title: Technology Knowledge Optimization in Type 1 Diabetes (TeKnO T1D): Parents
Acronym: TeKnO T1D
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the institution and is relinquishing the award supporting this study. The study will not launch.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-019791; K23DK129827 (NIH)
Record Dates: First submitted 2021-12-18; First posted 2022-03-29 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes
Keywords: pediatric; continuous glucose monitor; insulin pump; automated insulin delivery; hybrid closed loop systems; medical education; diabetes technology
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Semi-structured Interviews (No Intervention): Arm 1 will be conducted from months 0-15 and will use interviews to better understand existing challenges in diabetes technology educational practices. It is not a clinical trial, but is a crucial part of what builds to the clinical trial.
- Arm 2: Designing an App Delivered Curriculum (Experimental): Arm 2 will be conducted from months 10-33 and will use information learned in arm 1 to develop and beta test an educational curriculum. Arm 2 also is not a clinical trial, but is a crucial part of what builds to the clinical trial.
  Interventions: Other: TeKnO T1D: Parents
- Arm 3: TeKnO T1D: Parents Pilot Study (Active Comparator): Arm 3 will be conducted from months 30-60 and involves a pilot and feasibility study of the newly developed educational curriculum. This is the clinical trial.
  Interventions: Other: TeKnO T1D: Parents

INTERVENTIONS:
Other: TeKnO T1D: Parents — app-delivered curriculum to provide psychoeducational education surrounding diabetes technology use
  Arms: Arm 2: Designing an App Delivered Curriculum; Arm 3: TeKnO T1D: Parents Pilot Study

SUMMARY:
This study aims to identify the unmet psychoeducational needs of parents of children 8-12 years of age using insulin pump and CGM for pediatric T1D management and to leverage that information to develop an innovative app-based psychoeducational intervention to optimize use of these technologies and improve T1D outcomes.

DETAILED DESCRIPTION:
Despite increased use of insulin pumps and continuous glucose monitors (CGM) for pediatric type 1 diabetes (T1D) management and research studies showing benefits from the use of these devices, real-world glycemic control among youth with T1D has worsened in recent years. Although greater youth and parental diabetes knowledge is associated with better glycemic control, education alone is not sufficient to bring about the behavioral changes needed to improve outcomes in T1D. Psychoeducation recognizes the need to blend educational and behavioral approaches, including problem-solving and goal-setting, to support parents in developing optimal T1D management approaches. There are currently a lack of effective standardized tools to support patients and families in developing the knowledge and behavioral strategies needed to optimize the use of diabetes technologies. The development of innovative family-centered psychoeducational tools addressing both behavior and knowledge will help to realize the full potential of diabetes technologies to improve glycemic control and quality of life while ultimately preventing or delaying the development of both acute and long-term complications of T1D.

Interviews with parent-child dyads and diabetes clinicians will be used to identify the unmet parental psychoeducational needs regarding insulin pumps and CGM. These results will inform the use of instructional design to adapt an existing app-delivered diabetes technology curriculum to meet the specific needs of parents of children with T1D. Finally, the investigators will assess the feasibility and acceptability of this novel family-facing psychoeducational app-delivered intervention in a non-randomized pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. child 8-12 years of age with a diagnosis of T1D ≥ 6 months
2. currently using insulin pump( IP) and CGM ≥ 1 month [including Hybrid Closed Loop (HCL) systems]
3. participation of primary diabetes caregiver
4. English fluency
5. mean A1c >7.5% over the past 6 months (Aim 3 only)

Exclusion Criteria:

1. major illnesses other than T1D in the child
2. significant cognitive limitations or major psychiatric disorders in the child or parent
3. the use of medications other than insulin to control blood glucose levels.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Study Recruitment | Arm 3: Months 30-60
  Percentage of eligible patients who are approached and enroll in the study in Arm 3.
Intervention Satisfaction | Arm 3: Months 30-60
  Score on a survey developed to assess satisfaction with the Technology Knowledge Optimization Type 1 Diabetes: Parents curriculum in Arm 3. Scores range from 0-100 with higher scores reflecting greater satisfaction.
Perceived Intervention Utility | Arm 3: Months 30-60
  Score on a survey developed to assess the perceived utility of the Technology Knowledge Optimization Type 1 Diabetes: Parents curriculum during Arm 3. Scores range from 0-100 with higher scores reflecting greater perceived utility.
Intervention Completion | Arm 3: Months 30-60
  Percentage of enrolled participants who complete the TeKnO T1D: Parents Curriculum in Arm 3.
Intervention Retention | Arm 3: Months 30-60
  Percentage of enrolled participants who complete the entire intervention for Arm 3.

SECONDARY OUTCOMES:
Hemoglobin A1c | Arm 3: Months 30-60
  Hemoglobin A1c will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
CGM Mean Sensor Glucose | months 0-60
  CGM mean sensor glucose will be assessed prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
CGM Glucose Management Indicator | Arm 3: Months 30-60
  The Glucose Management Indicator will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
CGM Coefficient of Variation of the Mean | Arm 3: Months 30-60
  The Coefficient of Variation of the Mean will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. .
CGM Time in Range (70-180 mg/dL) | Arm 3: Months 30-60
  CGM Time in Range (70-180 mg/dL) will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
CGM Time Below Range (<70 mg/dL) | Arm 3: Months 30-60
  CGM Time Below Range (<70 mg/dL) will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
CGM Time Above Range (<180 mg/dL) | Arm 3: Months 30-60
  CGM Time Above Range (<180 mg/dL) will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
CGM Wear Time | Arm 3: Months 30-60
  The percentage of CGM wear time will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Total Daily Insulin Dose | Arm 3: Months 30-60
  Total Daily Insulin Dose will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Total Daily Basal Insulin Dose | Arm 3: Months 30-60
  Total Daily Basal Insulin Dose will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Percent Basal Insulin Dose | Arm 3: Months 30-60
  The percentage of the total daily insulin derived from basal insulin (basal insulin/ total daily insulin dose) will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Number of boluses per day | Arm 3: Months 30-60
  The number of boluses per day will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Carbohydrate intake logged on insulin pump | Arm 3: Months 30-60
  The number of grams of carbohydrate intake logged on insulin pump will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Episodes of Severe Hypoglycemia | Arm 3: Months 30-60
  The number of episodes of severe hypoglycemia will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Emergency Department Visits | Arm 3: Months 30-60
  The number of diabetes-related emergency department visits will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Hospital Admissions | Arm 3: Months 30-60
  The number of diabetes-related hospital admissions will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Episodes of Diabetic Ketoacidosis | Arm 3: Months 30-60
  The number of episodes of diabetic ketoacidosis will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Parent Diabetes-Specific Quality of Life | Arm 3: Months 30-60
  The Type 1 Diabetes and Life (T1DAL) is a validated survey assessing diabetes-specific quality of life. T1DAL will be will be completed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. Scores range from 0 to 100 with higher scores reflecting greater quality of life.
Parent Emotional Distress Related to T1D | Arm 3: Months 30-60
  Parents of Children (P-PAID) is a validated survey assessing emotional distress related to T1D. P-PAID will be completed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. Scores range from 15 to 96 with higher scores reflecting greater emotional distress.
Parent Diabetes Self-Management | Arm 3: Months 30-60
  The Diabetes Management Questionnaire (DMQ) is a validated survey assessing diabetes self-management. The DMQ will be completed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. Scores range from 0 to 100 with higher scores reflecting greater adherence to diabetes management.
Parent Perceived CGM Benefits and Burdens | months 0-60
  CGM Benefits and Burdens scale is a validated survey exploring perceived benefits and burdens of CGM use. CGM Benefits and Burdens will be completed prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. Scoring of the CGM Benefits subscale ranges from 1 to 40 with higher scores reflecting greater perceived benefits. Scoring of the CGM Burdens subscale ranges from 1 to 40 with higher scores reflecting less perceived burden.
Parent Diabetes Technology Knowledge | Arm 3: Months 30-60
  A survey assessing diabetes technology knowledge will be developed. This survey will be completed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. Scores range from 0 to 100 with higher scores reflecting greater knowledge.
Child Diabetes-Specific Quality of Life | Arm 3: Months 30-60
  The Type 1 Diabetes and Life (T1DAL) is a validated survey assessing diabetes-specific quality of life. T1DAL will be completed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. Scores range from 0 to 100 with higher scores reflecting greater quality of life.
Child Emotional Distress Related to T1D | Arm 3: Months 30-60
  Problem Areas in Diabetes- Child Version (PAID-C) is a validated survey assessing emotional distress related to T1D. PAID-C will be completed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion). Scores range from 11 to 84 with higher scores reflecting greater emotional distress.
Child Diabetes Self-Management | Arm 3: Months 30-60
  The Diabetes Management Questionnaire (DMQ) is a validated survey assessing diabetes self-management. The DMQ will be completed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. Scores range from 0 to 100 with higher scores reflecting greater adherence to diabetes management.
Child Perceived CGM Benefits and Burdens | Arm 3: Months 30-60
  CGM Benefits and Burdens scale is a validated survey exploring perceived benefits and burdens of CGM use. CGM Benefits and Burdens will be completed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion. Scoring of the CGM Benefits subscale ranges from 1 to 40 with higher scores reflecting greater perceived benefits. Scoring of the CGM Burdens subscale ranges from 1 to 40 with higher scores reflecting less perceived burden.

OTHER OUTCOMES:
Qualitative analysis of semi-structured interviews | Arm 1: Months 0-15
  Semantic content analysis will identify widely captured themes pertaining to diabetes technology education so as to prioritize content to include in curriculum development.
TeKnO T1D: Parents Curriculum difficulty | Arm 2: Months 10-33
  Using classical test theory as our framework, the investigators will conduct an item analysis to assess the quality of the items and the overall test, including item difficulty.
TeKnO T1D: Parents Curriculum discrimination | Arm 2: Months 10-33
  Using classical test theory as our framework, the investigators will conduct an item analysis to assess the quality of the items and the overall test, including item discrimination.
Child Weight Z-score | Arm 3: Months 30-60
  Weight Z-score for age will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Child Height Z-score | Arm 3: Months 30-60
  Height Z-score for age will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.
Child BMI Z-score | Arm 3: Months 30-60
  BMI Z-score for age will be assessed in Arm 3 prior to the curriculum start, upon completion of the TeKnO T1D: Parents curriculum, and 12 weeks after the curriculum completion.

CONTACTS AND LOCATIONS:
Overall Officials: Brynn E Marks, MD, MSHPEd, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No